CLINICAL TRIAL: NCT03292588
Title: Mechanisms Underlying Asthma Exacerbations Prevented and Persistent With Immune-Based Therapy: A Systems Approach Phase 2 (ICAC-30)
Brief Title: A Trial of Mepolizumab Adjunctive Therapy for the Prevention of Asthma Exacerbations in Urban Children
Acronym: MUPPITS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network); GlaxoSmithKline (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ICAC-30; UM1AI114271 (NIH); NIAID CRMS ID#: 38189 (Other: DAIT NIAID)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Asthma
Keywords: urban setting; children and adolescents; double-masked, placebo-controlled randomized trial; asthma exacerbations (attacks); mepolizumab adjunctive therapy; asthma exacerbations prevention; difficult-to-control exacerbation-prone asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab; Interleukin-5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepolizumab (Experimental): Intervention: Mepolizumab plus guidelines-based standard of care asthma treatment.
  Interventions: Biological: Mepolizumab
- Placebo (Placebo Comparator): Intervention: Placebo for mepolizumab plus guidelines-based standard of care asthma treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab administered every 4 weeks by subcutaneous injection at a dose of:
  * 100 mg for participants ≥12 years of age and
  * 40 mg for participants ages 6 to 11 years and weighing ≥40 kg.
  Note: Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in the study under previous versions of the protocol and were initially assigned a 100 mg dose will have their dose reduced to 40 mg.
  Participants 11 years of age will increase to the 100 mg dose if they become age 12 years during the study.
  Other Names: Nucala®; anti-Interleukin 5 (IL5) antagonist monoclonal antibody
  Arms: Mepolizumab
Drug: Placebo — Placebo administered every 4 weeks by subcutaneous injection at a dose of:
  * 100 mg for participants ≥12 years of age and
  * 40 mg for participants ages 6 to 11 years and weighing ≥40 kg.
  Note: Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in the study under previous versions of the protocol and were initially assigned a 100 mg dose will have their dose reduced to 40 mg.
  Participants 11 years of age will increase to the 100 mg dose if they become age 12 years during the study.
  Other Names: Placebo for Mepolizumab
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if treatment with a medication called Nucala® (mepolizumab), given along with standard asthma care, makes children less likely to have asthma attacks.

DETAILED DESCRIPTION:
Asthma is a growing problem, especially in children. It causes frequent wheezing, shortness of breath, chest tightness, and cough. Asthma attacks, or exacerbations, are problems for children with asthma.

The purpose of this study is to see if treatment with a medication called mepolizumab (Nucala®), given along with standard asthma care, makes children less likely to have asthma attacks. Mepolizumab is a new drug that is approved by the Food and Drug Administration (FDA) for use in children with asthma who are aged 12 years and older. Mepolizumab is given by injection. It is being studied by other researchers in children aged 6-11 years.

All participants will be prescribed standard asthma medications by a clinician who is trained in asthma care. Medications will include controller medications, a rescue medication, and a medication for severe asthma attacks (prednisone). The amount of medication that participants receive may be increased or decreased during the study based on their symptoms and breathing test results. Study clinicians will treat all participants according to the same guidelines. These treatment guidelines are based on recommendations from a group of national experts in asthma. This study has been designed this way so that all participants will have safe and effective standard asthma care.

In order to enroll in this study, participants must be willing to have their asthma managed by the study clinician during the entire study period. Participants must also be willing to bring study medications to all study visits.

This study will include up to 20 study visits. Participant involvement in the study will endure for approximately 1 year.

During the treatment period, participants will be placed in one of two treatment groups:

* Mepolizumab injection and guidelines-based asthma care or
* Placebo injection and guidelines-based asthma care.

Participants will not be able to choose which group they are assigned. This assignment is random and by chance, much like flipping a coin. Participants will not know if they are receiving mepolizumab or placebo. Investigators will compare the study results between the participants of each group.

ELIGIBILITY:
Inclusion Criteria:

Study applicant(s) that fulfill all of the inclusion criteria and none of the exclusion criteria are eligible for the study-

* Participant and/or parent guardian must be able to understand and provide informed consent and age-appropriate assent;
* Must have a primary place of residence in one of the pre-selected recruitment census tracts as outlined in the study's Manual of Procedures (MOP);
* Has had a diagnosis of asthma made >1 year prior to recruitment;

  --Those who received an asthma diagnosis by a clinician ≤1 year prior to recruitment must report that their respiratory symptoms were present for more than 1 year prior to recruitment.
* Has had ≥2 asthma exacerbations in the prior year (defined as a requirement for systemic corticosteroids and/or hospitalization);
* At Visit 0 (Screening), has the following requirement for asthma controller medication:

  * For those ages 6 to 11 years, treatments with at least fluticasone 250 mcg dry powder inhaler (DPI) one puff twice daily or its equivalent and,
  * For those ≥12 years of age, treatment with at least Advair 250/50 mcg dry powder inhaler (DPI), one puff twice daily or its equivalent.
* Has peripheral blood eosinophils ≥150 cells/µl obtained at Visit 0 (Screening) or in another Inner-City Asthma Consortium (ICAC) clinical research study within 6 months;
* Is able to perform spirometry at randomization (Visit for treatment assignment);
* Has documentation of current medical insurance with prescription coverage at randomization; and
* Has had varicella or the varicella vaccination.

Exclusion Criteria:

Individual(s) who meets any of the following criteria are not eligible for enrollment or randomization-

* Is not able or willing to give written informed consent or comply with the study protocol;
* Has concurrent (existing) medical problems that would require systemic corticosteroids or other immunomodulator treatments during the study;
* Is currently receiving immunotherapy;
* Is currently receiving treatment with omalizumab or has had omalizumab treatment within 6 months prior to planned participant randomization to treatment assignment;
* Is currently requiring greater than fluticasone 500 mcg administered twice daily plus a long-acting beta agonist (LABA) one puff twice daily or its equivalent, and/or

  --Individuals using oral corticosteroids daily or every other day for more than 14 days at the time of Visit 0 (Screening).
* Is currently pregnant or lactating, or plans to become pregnant during the time of study participation

  --Note: Females of child-bearing potential (post-menarche) must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral subcutaneous, mechanical, or surgical contraception).
* Has a known, pre-existing clinically important lung condition other than asthma;
* Has a current malignancy or previous history of cancer in remission for less than 12 months prior to randomization;
* Has known, pre-existing, unstable liver disease;
* Is a current smoker or has a smoking history of 10 or more pack years;
* Has a known immunodeficiency disease;
* Has other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, including eosinophilic granulomatosis with polyangiitis;
* Has a known, active pre-existing parasitic infestation or is undergoing treatment for a parasitic infestation

  --Note: Once the individual has been successfully treated, the interested study applicant may be reevaluated for study eligibility.
* Positive for use of investigational drugs within 4 weeks of randomization;
* Has a past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the study clinician,

  * May pose additional risks from participation in this study,
  * May interfere with the participant's ability to comply with study requirements, or
  * May impact the quality or interpretation of the data obtained from the study.
* In the event that the study applicant will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol;
* Has a known history of allergic reaction to previous biologic therapy for asthma; or
* Has had a life threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation or resulting in a hypoxic seizure.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 335 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Jackson, MD, Study Chair — University of Wisconsin, Madison; William W Busse, MD, Study Chair — University of Wisconsin, Madison
Locations (9):
- United States (9):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials will be made available upon completion of the trial.
Time Frame: After completion of the trial, within 24 months status post database lock.
Access Criteria: Registration is available for the Immunology Database and Analysis Portal (ImmPort) at: https://www.immport.org/registration. Submit a rationale for the purpose of requesting study data access.
  ImmPort is a long-term archive of clinical and mechanistic data, a National Institute of Allergy and Infectious Diseases Division of Allergy, Immunology and Transplantation (NIAID DAIT)-funded data repository. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort is provided by NIH-funded programs, other research organizations and individual scientists, ensuring these discoveries will be the foundation of future research.
URL: https://www.immport.org/home

REFERENCES:
- [Derived] Gaberino CL, Segnitz RM, Dill-McFarland KA, Bacharier LB, Calatroni A, Gill MA, Stokes J, Liu AH, Cohen RT, Kumar R, Lang A, Khurana Hershey GK, Sherenian MG, Zoratti EM, Teach SJ, Kattan M, Becker PM, Togias A, Busse WW, Jackson DJ, Altman MC. Mepolizumab alters gene regulatory networks of nasal airway type-2 and epithelial inflammation in urban children with asthma. Nat Commun. 2025 Sep 2;16(1):8191. doi: 10.1038/s41467-025-63629-2. PMID 40897727
- [Derived] Altman MC, Janczyk T, Murphy RC, Jayavelu ND, Calatroni A, Kattan M, Gill MA, Stokes J, Liu AH, Khurana Hershey GK, Sherenian M, Kumar R, Robison RG, Gruchalla RS, O'Connor GT, Zoratti EM, Teach SJ, Lynch SV, Dill-McFarland KA, Becker PM, Togias A, Gern JE, Bacharier LB, Busse WW, Jackson DJ; Inner City Asthma Consortium and Childhood Asthma in Urban Settings Network. Inflammatory Pathways in Residual Asthma Exacerbations Among Mepolizumab-Treated Urban Children: A Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2025 Sep 1;179(9):957-970. doi: 10.1001/jamapediatrics.2025.2044. PMID 40658400
- [Derived] Jackson DJ, Bacharier LB, Gergen PJ, Gagalis L, Calatroni A, Wellford S, Gill MA, Stokes J, Liu AH, Gruchalla RS, Cohen RT, Makhija M, Khurana Hershey GK, O'Connor GT, Pongracic JA, Sherenian MG, Rivera-Spoljaric K, Zoratti EM, Teach SJ, Kattan M, Dutmer CM, Kim H, Lamm C, Sheehan WJ, Segnitz RM, Dill-McFarland KA, Visness CM, Becker PM, Gern JE, Sorkness CA, Busse WW, Altman MC; US National Institute of Allergy and Infectious Disease's Inner City Asthma Consortium. Mepolizumab for urban children with exacerbation-prone eosinophilic asthma in the USA (MUPPITS-2): a randomised, double-blind, placebo-controlled, parallel-group trial. Lancet. 2022 Aug 13;400(10351):502-511. doi: 10.1016/S0140-6736(22)01198-9. PMID 35964610
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 335 people were enrolled in the study (signed a consent and were assigned a unique participant number). However, 45 participants dropped out before receiving treatment bringing the total to 290 participants who started treatment.
Groups:
- Mepolizumab: Intervention: Mepolizumab plus guidelines-based standard of care asthma treatment.
  Mepolizumab: Mepolizumab administered every 4 weeks by subcutaneous injection at a dose of:
  * 100 mg for participants ≥12 years of age and
  * 40 mg for participants ages 6 to 11 years and weighing ≥40 kg.
  Note: Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in the study under previous versions of the protocol and were initially assigned a 100 mg dose will have their dose reduced to 40 mg.
  Participants 11 years of age will increase to the 100 mg dose if they become age 12 years during the study.
- Placebo: Intervention: Placebo for mepolizumab plus guidelines-based standard of care asthma treatment.
  Placebo: Placebo administered every 4 weeks by subcutaneous injection at a dose of:
  * 100 mg for participants ≥12 years of age and
  * 40 mg for participants ages 6 to 11 years and weighing ≥40 kg.
  Note: Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in the study under previous versions of the protocol and were initially assigned a 100 mg dose will have their dose reduced to 40 mg.
  Participants 11 years of age will increase to the 100 mg dose if they become age 12 years during the study.
Period: Overall Study
Arm/Group | Mepolizumab | Placebo
Started | 146 | 144
Completed | 126 | 122
Not Completed | 20 | 22
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 12 | 16
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Move out of town | 1 | 0
Not completed — >3 bursts of systemic corticosteroids for asthma during treatment period (Starting Nov 2020) | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population with available data
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab | Placebo | Total
Number analyzed (Participants) | 146 | 144 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 146 | 144 | 290
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (2.87) | 10.8 (2.88) | 10.8 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 55 | 126
  Male | 75 | 89 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 37 | 72
  Not Hispanic or Latino | 111 | 107 | 218
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 146 | 144 | 290

OUTCOME MEASURES:

1. Primary Outcome: Number of Asthma Exacerbations During the Treatment Period
Description: Exacerbations were defined as a prescription of a course of systemic corticosteroids by a clinician, initiation of a course of systemic corticosteroids by a participant, or as a hospitalization for asthma. If a participant initiated and completed a course of systemic corticosteroids without clinician involvement, this course was counted only if the study clinician agreed the treatment was warranted, and it met the following dosage: the course for prednisone, prednisolone, or methylprednisolone was at least 20 mg daily dose for 3 of 5 consecutive days. The course for dexamethasone was at least a 10 mg single daily dose. If a corticosteroid burst for the treatment of an asthma exacerbation was prescribed by a non-ICAC clinician, it was counted regardless of dose.
Time Frame: Up to 12 months
Population: All participants who were randomized and received at least one dose of study treatment
Measure: Mean (Standard Error); unit: Exacerbations during treatment
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
Exacerbations during treatment | 0.96 (0.10) | 1.30 (0.13)
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Test type: Superiority — Negative binomial model for the rate of exacerbations in the first year. The model included an offset term to account for differential follow-up among participants. To account for adaptive randomization, the model was also adjusted for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (< or ≥400 cells/μl), BMI (< or ≥95th percentile for age), total serum IgE (< or ≥540 kUA/L) and treatment dose (40 mg or 100 mg); p = 0.027, Regression, Negative Binomial; Adjusted relative rate of exacerbations in the first year; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.56 to 0.96]

2. Secondary Outcome: Composite Asthma Severity Index (CASI)
Description: Composite Asthma Severity Index (CASI) scores included 5 domains: day symptoms and albuterol use, night symptoms and albuterol use, controller treatment, lung function measures, and exacerbations. The minimum composite score was 0 while the maximum was 20. The higher the score the more allergy symptoms a subject has.
Time Frame: Week 12, 24, 36, 48, 52 after randomization
Population: All participants who were randomized and received at least one dose of study treatment
Measure: Least Squares Mean (Standard Error); unit: Composite Asthma Severity Index
Groups:
- Mepolizumab: Mepolizumab (anti-IL-5 antagonist monoclonal antibody) by subcutaneous injection every 4 weeks at the following doses: Age 12 years and above-100 mg, Age 6-11 years-40mg, Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in Protocol ICAC-30 under the previous versions of the protocol and initially assigned a 100 mg dose will have their dose reduced to 40 mg
- Placebo: Placebo by subcutaneous injection every 4 weeks at the following doses: Age 12 years and above-100 mg, Age 6-11 years-40mg, Participants 6 to 11 years of age and weighing ≥40 kg who were enrolled in Protocol ICAC-30 under the previous versions of the protocol and initially assigned a 100 mg dose will have their dose reduced to 40 mg
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
Composite Asthma Severity Index
  Week 12 | 6.17 (0.2) | 6.45 (0.20)
  Week 24 | 5.94 (0.23) | 6.01 (0.23)
  Week 36 | 5.48 (0.22) | 5.99 (0.23)
  Week 48 | 5.16 (0.22) | 5.23 (0.22)
  Week 52 | 5.03 (0.23) | 5.00 (0.23)
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Week 12; Test type: Superiority; p = 0.290, Mixed Models Analysis; The difference in least square mean of CASI scores for week 12; Least Square Mean Difference = -0.28, 95% CI 2-sided [-0.81 to 0.24]
Statistical Analysis 2: Comparison: Mepolizumab vs Placebo; Week 24; Test type: Superiority; p = 0.820, Mixed Models Analysis; The difference in least square mean of CASI scores for week 24; Least Square Mean Difference = -0.07, 95% CI 2-sided [-0.69 to 0.55]
Statistical Analysis 3: Comparison: Mepolizumab vs Placebo; Week 36; Test type: Superiority; p = 0.096, Mixed Models Analysis; The difference in least square mean of CASI scores for week 36; Least Square Mean Difference = -0.51, 95% CI 2-sided [-1.11 to 0.09]
Statistical Analysis 4: Comparison: Mepolizumab vs Placebo; Week 48; Test type: Superiority; p = 0.831, Mixed Models Analysis; The difference in least square mean of CASI scores for week 48; Least Square Mean Difference = -0.06, 95% CI 2-sided [-0.65 to 0.52]
Statistical Analysis 5: Comparison: Mepolizumab vs Placebo; Week 52; Test type: Superiority; p = 0.947, Mixed Models Analysis; The difference in least square mean of CASI scores for week 52; Least Square Mean Difference = 0.02, 95% CI 2-sided [-0.60 to 0.64]

3. Secondary Outcome: Participant Quality of Life Measured Using the Physician Global Assessment Tool
Description: The Physician Global Assessment Tool was used to assess the quality of life of the subjects during treatment. The questionnaire is one question that asks the physician to evaluate how the participant's quality of life changed over the course of treatment. There are seven possible options ranging from significantly worse to significantly improved.
Time Frame: Week 56
Population: All participants who were randomized and received at least one dose of study treatment and completed the quality of life questionnaire at visit 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 129 | 122
Participants
  Physician Global Assessment Tool - Significantly Improved | 58 | 54
  Physician Global Assessment Tool - Moderately Improved | 27 | 33
  Physician Global Assessment Tool - Mildly Improved | 22 | 17
  Physician Global Assessment Tool - No Change | 20 | 17
  Physician Global Assessment Tool - Mildly Worse | 1 | 1
  Physician Global Assessment Tool - Moderately Worse | 0 | 0
  Physician Global Assessment Tool - Significantly Worse | 1 | 0
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Physician Global Assessment Tool; Test type: Superiority — A generalized logit model was used to analyze Physician Global Assessment Tool at Visit 14. The model included treatment arm as fixed effect as primary exposure but was also adjusted for study site, # of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils ((< or ≥400 cells/μl), BMI (< or ≥95th percentile for age) & total serum IgE (< or ≥540 kUA/L). No imputation of missing data was used for participants who weren't assessed for quality of life measurements at Visit 14; p = 0.974, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.62 to 1.64]

4. Secondary Outcome: Participant Quality of Life Measured Using the Patient Global Assessment, at Visit 14
Description: The Patient Global Assessment Tool was used to assess the quality of life of the subjects during treatment. The questionnaire is one question that asks the participant to evaluate how their quality of life changed over the course of treatment. There are seven possible options ranging from significantly worse to significantly improved.
Time Frame: Week 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 129 | 124
Participants
  Patient Global Assessment Tool - Significantly Improved | 82 | 87
  Patient Global Assessment Tool - Moderately Improved | 27 | 23
  Patient Global Assessment Tool - Mildly Improved | 11 | 12
  Patient Global Assessment Tool - No Change | 7 | 2
  Patient Global Assessment Tool - Mildly Worse | 2 | 0
  Patient Global Assessment Tool - Moderately Worse | 0 | 0
  Patient Global Assessment Tool - Significantly Worse | 0 | 0
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Patient Global Assessment Tool; Test type: Superiority — A generalized logit model was used to analyze the Patient Global Assessment Tool at Visit 14. The model included treatment arm as fixed effect as the primary exposure but was adjusted for study site, # of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils ((< or ≥400 cells/μl), BMI (< or ≥95th percentile for age) & total serum IgE (< or ≥540 kUA/L). No imputation of missing data was used for participants who weren't assessed for quality of life measurements at Visit 14; p = 0.238, Regression, Logistic; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.42 to 1.24]

5. Secondary Outcome: Lung Function as Assessed by Spirometry
Description: A generalized mixed model was used to analyze spirometry parameter at each visit where the lung function was collected. The ratio of the forced expiratory volume to the forced vital capacity of the lungs (FEV1/FVC) is the outcome that measured lung function.
Time Frame: Weeks 12, 24, 36, 48, 52 after randomization
Population: All participants who were randomized and received at least one dose of study treatment
Measure: Least Squares Mean (Standard Error); unit: FEV1/FVC
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
FEV1/FVC
  FEV1/FVC - Week 12 | 0.747 (0.007) | 0.752 (0.007)
  FEV1/FVC - Week 24 | 0.755 (0.007) | 0.766 (0.007)
  FEV1/FVC - Week 36 | 0.758 (0.008) | 0.747 (0.008)
  FEV1/FVC - Week 48 | 0.755 (0.008) | 0.742 (0.008)
  FEV1/FVC - Week 52 | 0.761 (0.008) | 0.763 (0.008)
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; FEV1/FVC Week 12; Test type: Superiority — A generalized mixed model as described in section 8.3.1 was used to analyze each spirometry and impulse oscillometry parameter, separately, at each visit where the lung function was collected; p = 0.591, Mixed Models Analysis; Least Square Mean Difference = -0.005, 95% CI 2-sided [-0.023 to 0.013]
Statistical Analysis 2: Comparison: Mepolizumab vs Placebo; FEV1/FVC Week 24; Test type: Superiority; p = 0.265, Mixed Models Analysis; Least Square Mean Difference = -0.011, 95% CI 2-sided [-0.031 to 0.008]
Statistical Analysis 3: Comparison: Mepolizumab vs Placebo; FEV1/FVC Week 36; Test type: Superiority; p = 0.345, Mixed Models Analysis; Least Square Mean Difference = 0.011, 95% CI 2-sided [-0.012 to 0.033]
Statistical Analysis 4: Comparison: Mepolizumab vs Placebo; FEV1/FVC Week 48; Test type: Superiority; p = 0.248, Mixed Models Analysis; Least Square Mean Difference = 0.013, 95% CI 2-sided [-0.009 to 0.036]
Statistical Analysis 5: Comparison: Mepolizumab vs Placebo; FEV1/FVC Week 52; Test type: Superiority; p = 0.864, Mixed Models Analysis; Least Square Mean Difference = -0.002, 95% CI 2-sided [-0.023 to 0.020]

6. Secondary Outcome: Lung Function as Assessed by Impulse Oscillometry
Description: A generalized mixed model was used to analyze impulse oscillometry parameter at each visit where the lung function was collected. The Percent Predicted FEV1 (%) is the outcome that measured lung function.
Time Frame: Weeks 12, 24, 36, 48, 52 after randomization
Measure: Least Squares Mean (Standard Error); unit: Percent Predicted FEV1 (%)
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
Percent Predicted FEV1 (%)
  FEV1PP - Week 12 | 91.9 (1.27) | 92.3 (1.27)
  FEV1PP - Week 24 | 90.8 (1.46) | 94.2 (1.49)
  FEV1PP - Week 36 | 91.5 (1.45) | 89.9 (1.46)
  FEV1PP - Week 48 | 90.4 (1.46) | 89.8 (1.48)
  FEV1PP - Week 52 | 90.9 (1.45) | 93.5 (1.43)
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; FEV1PP Week 12; Test type: Superiority; p = 0.816, Mixed Models Analysis; Least Square Mean Difference = -0.4, 95% CI 2-sided [-3.8 to 3.0]
Statistical Analysis 2: Comparison: Mepolizumab vs Placebo; FEV1PP Week 24; Test type: Superiority; p = 0.095, Mixed Models Analysis; Least Square Mean Difference = -3.4, 95% CI 2-sided [-7.4 to 0.6]
Statistical Analysis 3: Comparison: Mepolizumab vs Placebo; FEV1PP Week 36; Test type: Superiority; p = 0.444, Mixed Models Analysis; Least Square Mean Difference = 1.5, 95% CI 2-sided [-2.4 to 5.5]
Statistical Analysis 4: Comparison: Mepolizumab vs Placebo; FEV1PP Week 48; Test type: Superiority; p = 0.751, Mixed Models Analysis; Least Square Mean Difference = 0.6, 95% CI 2-sided [-3.3 to 4.6]
Statistical Analysis 5: Comparison: Mepolizumab vs Placebo; FEV1PP Week 52; Test type: Superiority; p = 0.184, Mixed Models Analysis; Least Square Mean Difference = -2.6, 95% CI 2-sided [-6.5 to 1.3]

7. Secondary Outcome: Rate of Exacerbations (Mepolizumab vs. Placebo) During the Treatment Period for Participants Who Did Not Fit the FDA-approved Dosing Table for Omalizumab Therapy.
Description: Looking at the rate of exacerbations similarly to the primary endpoint. This outcome measure also took into consideration FDA- approved dosing of omalizumab. The FDA-approved dosing table is based off of age, weight and pre-treatment Serum IGE
Time Frame: Up to 12 months
Measure: Mean (Standard Error); unit: Exacerbations during treatment
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 57 | 51
Exacerbations during treatment | 1.11 (0.21) | 1.31 (0.25)
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Did not meet FDA-approved dosing; Test type: Superiority — Negative binomial model for the rate of exacerbations (per year. The model included an offset term to account for differential follow-up among participants. To account for adaptive randomization, the model was also adjusted for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (< or ≥400 cells/μl), BMI (< or ≥95th percentile for age), total serum IgE (< or ≥540 kUA/L) and treatment dose (40 mg or 100 mg); p = 0.458, Mixed Models Analysis; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.55 to 1.31]

8. Secondary Outcome: Rate of Exacerbations (Mepolizumab vs. Placebo) During the Treatment Period for Participants Who Fit the FDA-approved Dosing Table.
Description: as for outcome 7
Time Frame: Up to 12 months
Measure: Mean (Standard Error); unit: Exacerbations during treatment
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 89 | 93
Exacerbations during treatment | 0.87 (0.13) | 1.30 (0.18)
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Fit FDA-approved dosing; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.025, Regression, Negative Binomial; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.47 to 0.95]

9. Secondary Outcome: Time to First Asthma Exacerbation
Description: A Cox PH model was also used to model the time to first asthma exacerbation during the treatment period. The Cox PH model included treatment arm as the primary exposure but was also adjusted for study site, number of exacerbations in year prior to study (2 or 3+), peripheral blood eosinophils (above or below 400 cells/μl), BMI (above or below 95th percentile for age) and total serum IgE (above or below 540 kUA/L).
Time Frame: Up to 12 months
Population: All participants who were randomized and received at least one dose of study treatment
Measure: Median (Full Range); unit: Days
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
Days | 241 [1 to 380] | 224 [1 to 378]
Statistical Analysis 1: Comparison: Mepolizumab vs Placebo; Test type: Superiority; p = 0.3587, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.63 to 1.18]

10. Secondary Outcome: Number of Reported Adverse Events (AEs), Including Their Severity
Description: The number of AEs by severity was used to assess safety. Please refer to the Adverse Event tables for specifics.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Population: Number of Subjects with at Least One AE by severity
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 113 | 94
Participants
  Severity: Grade 1 - Mild | 47 | 39
  Severity: Grade 2 - Moderate | 58 | 51
  Severity: Grade 3 - Severe and undesirable | 8 | 3
  Severity: Grade 4 - Life-threatening or disabling | 0 | 1
  Severity: Grade 5 - Death | 0 | 0

11. Secondary Outcome: Number of Reported Adverse Events (AEs), Including Their Treatment Relatedness
Description: The number of AEs by relationship to study drug was used to assess safety. Please refer to the Adverse Event tables for specifics.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Population: Number of Subjects with any study procedures related AEs
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
Participants | 46 | 26

12. Secondary Outcome: Number of Reported Serious Adverse Events (SAEs) Inclusive of Severity. Please Refer to the Adverse Event Tables for Specifics.
Description: The number of SAEs by severity and relationship to study drug was used to assess safety.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Population: Number of subjects with Serious Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 4 | 2
Participants
  Severity: Grade 2 - Moderate | 0 | 1
  Severity: Grade 3 - Severe and undesirable | 3 | 1
  Severity: Grade 4 - Life threatening | 0 | 0
  Severity: Grade 5 - Death | 1 | 0

13. Other Pre Specified Outcome: EXPLORATORY: Time to First Respiratory Virus-Induced Exacerbation
Description: As measured by an exacerbation associated with a respiratory virus detected using nasal mucus samples obtained at the time of an exacerbation.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: EXPLORATORY:Number of Respiratory Virus-Induced Exacerbations
Description: Measured by an exacerbation associated with a respiratory virus detected using nasal mucus samples obtained at the time of an exacerbation.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: EXPLORATORY:Childhood Asthma Control Test (ACT)/c-ACT
Description: A validated tool to assess overall asthma control (over the last 4 weeks) in participants.
Time Frame: Visits (V) 4 (Week 4 Treatment Initiation) , V4 (Week 16), V7 (Week 28), V10 (Week 40), V13 (Week 52) and V14 (Week 56, Completion of Treatment)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: EXPLORATORY:Maximum Number of Asthma Symptom Days
Description: Defined as the highest value among the following variables over a two-week period:
  * number of days with wheezing, tightness in the chest, or cough;
  * number of nights with disturbed sleep as a result of asthma; and
  * number of days on which the participant had to slow down or discontinue play/physical activities.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: EXPLORATORY:Bronchodilator Responsiveness
Description: A measure to determine whether mepolizumab improves pulmonary outcomes.
Time Frame: Baseline (prior to treatment initiation), Week 56 (Completion of Treatment)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: EXPLORATORY: Gene Expression in Nasal Lavage Samples
Description: Whole genome transcriptomics of nasal lavage samples to identify inflammatory pathways affected by mepolizumab.
Time Frame: Visits (V) 1 (Week 4 Treatment Initiation) , V3(Week 12), and V14 (Week 56, Completion of Treatment)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: EXPLORATORY: Gene Expression in Whole Blood RNA Samples
Description: Whole genome transcriptomics of whole blood RNA samples to identify inflammatory pathways affected by mepolizumab..
Time Frame: Visits (V) 1 (Week 4 Treatment Initiation) , V3(Week 12), and V14 (Week 56, Completion of Treatment)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: EXPLORATORY:Levels of Antibody to Mepolizumab
Description: An assay for detection/measurement of levels of antibody to mepolizumab. Analysis will include participants randomized to mepolizumab.
Time Frame: Visit (V) 1 (Week 4, prior to treatment initiation), V3 (Week 12), and Visit 14 (Week 56, Completion of Treatment)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: EXPLORATORY:Other Potential Biomarkers Not Specified to Date
Description: Plasma, nasal samples, RNA and DNA will be banked for possible future study of potential biomarkers associated with asthma and asthma exacerbations.
Time Frame: Visit (V) 1 (Week 4, prior to treatment initiation), V3 (Week 12), and Visit 14 (Week 56, Completion of Treatment)
Reporting Status: Not Posted

22. Secondary Outcome: Number of Reported Serious Adverse Events (SAEs) Inclusive of Treatment Relatedness. Please Refer to the Adverse Event Tables for Specifics.
Description: The number of SAEs by relationship to study drug was used to assess safety.
Time Frame: Week 4 (Treatment Initiation) to Week 56 (Completion of Treatment)
Population: Number of subjects with any study procedures related Serious Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab | Placebo
Number analyzed (Participants) | 146 | 144
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until 1 year and the participant completes study participation or until 30 days after he/she prematurely withdraws (without withdrawing consent) or is withdrawn from the study.
Description: The safety population was used for reporting adverse events, which was defined as: participants who were randomized and received at least one dose of study treatment. Participants were analyzed according to the medication they actually received, regardless of the treatment arm to which they were randomized. Non-treatment emergent adverse events were summarized in all participants who were enrolled, while treatment emergent adverse events were summarized in the safety sample
Arm/Group | Mepolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/146 | 0/144
Serious Adverse Events (participants affected / at risk) | 4/146 | 2/144
Other Adverse Events (participants affected / at risk) | 53/146 | 42/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab (N=146) | Placebo (N=144)
All-Cause Mortality (General disorders) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab (N=146) | Placebo (N=144)
Vomiting (Gastrointestinal disorders) | 13 (15) | 12 (13)
Injection site reaction (General disorders) | 13 (14) | 0 (0)
Influenza (Infections and infestations) | 11 (11) | 11 (11)
Pharyngitis streptococcal (Infections and infestations) | 7 (7) | 9 (9)
Headache (Nervous system disorders) | 15 (19) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03292588/Prot_SAP_000.pdf